CLINICAL TRIAL: NCT04724291
Title: Magnetically Controlled Capsule for Assessment of Gastric Mucosa in Symptomatic Patients
Brief Title: MAGNET (Magnetically Controlled Capsule for Assessment of Gastric Mucosa in Symptomatic Patients)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Andrew Meltzer, Associate Professor of Medicine, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCR191848
Record Dates: First submitted 2020-10-01; First posted 2021-01-26 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Pain; Gastritis; Gastric Ulcer; Gastric Cancer
Keywords: capsule endoscopy; EGD
MeSH Terms: conditions — Abdominal Pain; Gastritis; Stomach Ulcer; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MAGNET + EGD (Other): Capsule endoscopy followed by traditional endoscopy
  Interventions: Device: MAGNET

INTERVENTIONS:
Device: MAGNET — This study will test the accuracy of a single-use ingestible video capsule (NaviCamTM, AnX Robotica) which is remotely controlled to record images of the inside of your stomach. Participants in this research study will have symptoms for which an evaluation by a traditional tube-based endoscopy (EGD) is indicated.

SUMMARY:
This pilot and feasibility study will be first US study to determine if a magnetically controlled capsule (MCC) can effectively visualize the anatomy of the stomach like a more traditional upper endoscopy (EGD). This study is designed to enroll participants who have a standard indication for an EGD and are also willing to get an MCC exam. The MCC is driven actively by a clinician unlike prior capsule endoscopes that move passively by gravity or peristalsis. Thus, a physician will be able to look more closely at areas of the stomach that might be concerning and might need further evaluation and/or treatment.

DETAILED DESCRIPTION:
In the United States, upper endoscopy is frequently performed for a variety of symptoms including heartburn, bloating, nausea, burping, and epigastric pain/burning. The prevalence of these symptoms may provide as much as 25% of a gastroenterologist's office practice. In general, the diagnostic yield of an EGD is low. Without alarm symptoms, as many as 70% of procedures are negative for significant findings. One major indication is testing for H. pylori for which EGD may be unnecessary, because H. pylori detection can be accomplished by fecal antigen testing or breath testing as accurately as biopsy and less expensively.

Investigators believe there is an opportunity to improve the risk stratification of patients that undergo endoscopy through the use of MCC. Our primary hypothesis is that MCC allows for visualization of the stomach of symptomatic patients referred from the emergency department, urgent care, and primary care settings with clinical symptoms appropriate for endoscopy. A prospective study is proposed to evaluate the feasibility, safety and accuracy of this novel diagnostic modality.

Esophagogastroduodenoscopy (EGD) is one of the most common medical procedures and indications for epigastric pain, bloating, burning, heart-burn, excessive belching, nausea, vomiting, anemia, and weight loss. Access to EGD is limited by the cost, the need for an endoscopy specialist and the need for anesthesia. Lack of access to an EGD is a health disparity associated with increased gastric cancer mortality-to-incidence ratio. A novel approach to visualization of the upper GI tract is needed to increase access to care and improve diagnostic capabilities. Magnetically controlled capsule (MCC) is the first wireless ingestible capsule endoscope that is able to be directed by operator to visualize all anatomic areas of the stomach (NaviCam™, AnX Robotica). This study will be the first US study to examine the feasibility of using MCC in patients with relevant symptoms to the stomach. The goal is to ascertain if the diagnostic capabilities of the MCC compared to EGD are comparable for symptomatic patients who have clinical indications for an EGD.

MCC offers potential advantages over traditional EGD including the ability to be performed 24 hours a day without sedation and to be performed without an endoscopist. In addition, the MCC is less invasive, does not cause discomfort, and enables the patient to pursue normal daily activities after the procedure. Non-specialist physicians can administer the MCC and interpretation can be done in real-time or asynchronously by GI specialists. The MCC may impact decisions regarding the need for hospitalization, the need for additional diagnostic testing such as biopsy, the need for additional therapeutic interventions such as endoscopic hemostasis and polypectomy, and the need for further risk stratification of disease. The eventual work-flow may be similar to that of many current diagnostic tests such as radiologic examinations. This ability to transmit images could become especially important in rural communities or in communities that have limited access to a gastroenterologist or surgeon. Incorporation of the MCC into current practice could follow a trajectory similar to that of point-of-care ultrasonography, an imaging modality in which non-radiologist physicians have become increasingly skilled and for which indications continue to expand. The American Society of Gastrointestinal Endoscopy states that credentials for capsule endoscopy should be determined independently from other endoscopic procedures such as colonoscopy, sigmoidoscopy, or any other endoscopic procedure. The American Society of Gastrointestinal Endoscopy also emphasizes sound medical training, appropriate patient selection, correct interpretation, and continued medical management for these capsule endoscopists. Capsule endoscopy requires only image interpretation and does not require procedural skill training associated with other endoscopic procedures; therefore, ED physicians, urgent care physicians, primary care doctors, and mid-level practitioners can meet these criteria with basic training.

Contraindications to the MCC are similar to contraindications for established capsule endoscopy (CE) which has been performed safely in a variety of clinical settings. The only absolute contraindication is intestinal obstruction. There is a low risk of non-natural excretion of capsules estimated at less than 1 in 100. In general, the CE procedure poses significantly less risk than traditional EGD, and multiple studies have shown that CE is well tolerated in patients with acute symptoms.

The cost of the capsule is an important factor that may affect future use in the ED and clinics. The use of MCC in the ED, urgent care and primary care can potentially lead to more patients being safely managed in an outpatient setting. MCC may be especially cost-effective if it reduces hospital admissions, need for anesthesia, missed work days or overall EGDs. Future technological developments in the MCC may allow for operator to collect biopsy samples and perform therapeutic functions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥ 18 years with upper GI symptoms (epigastric pain/burning, bloating, heart-burn, excessive belching, nausea/vomiting, anemia, and/or weight loss) appropriate for an upper endoscopy evaluation
* Able to speak English
* Able to understand and sign consent form
* Able to undergo standard outpatient endoscopy
* Indications for traditional EGD in the next 30 days

  * Low blood (Unexplained anemia)
  * Blood in vomit (Hematemesis)
  * Upper abdominal or chest pain
  * Indigestion (Dyspepsia)
  * GERD
  * Suspected ulcers
  * Unexplained weight loss
  * Gastric Biopsy
  * Other

Exclusion Criteria:

* Hemodynamic shock
* Active hematemesis
* Dysphagia, swallowing disorder, Zenker's diverticulum, suspected bowel obstruction or perforation, gastroparesis, gastric outlet obstruction, Crohn's disease, prior GI tract surgery that changes the gastrointestinal anatomy (e.g., Billroth I or II, esophagectomy, gastrectomy, bariatric procedure and small intestinal resection)
* Presumed pregnant, trying to conceive or currently breastfeeding
* Altered mental status (e.g., hepatic encephalopathy) that limits the ability to swallow a capsule
* Expected to have Magnetic Resonance Imaging examination within 30 days
* Currently (<12 hours) on medications that may coat the upper GI tract such as antacids or sucralfate or Maalox
* No reliable contact information--no phone, no permanent address
* ASA status of more than 3
* Implanted with a cardiac pacemaker or other implantable electronic medical device
* BMI is greater than or equal to 38

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Meltzer, MD, MS, Principal Investigator — George Washington University; Anita Kumar, MD, Principal Investigator — George Washington University; Marie Borum, MD, Principal Investigator — George Washington University; Samuel Schueler, MD, Principal Investigator — George Washington University; David Cave, MD, Principal Investigator — UMass Memorial Health; Samuel J Kallus, MD, Principal Investigator — George Washington University School of Medicine and Health Sciences
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White CM, Kilgore ML. PillCam ESO versus esophagogastroduodenoscopy in esophageal variceal screening: A decision analysis. J Clin Gastroenterol. 2009 Nov-Dec;43(10):975-81. doi: 10.1097/MCG.0b013e3181a7ed09. PMID 19661814
- [Background] Seddighzadeh A, Wolf AT, Parasuraman S, Shetty R, Vallurupalli N, Reddy S, Goldhaber SZ. Gastrointestinal complications after 3 months of dual antiplatelet therapy for drug-eluting stents as assessed by wireless capsule endoscopy. Clin Appl Thromb Hemost. 2009 Mar-Apr;15(2):171-6. doi: 10.1177/1076029608325545. Epub 2008 Dec 30. PMID 19117963
- [Background] Gralnek IM, Adler SN, Yassin K, Koslowsky B, Metzger Y, Eliakim R. Detecting esophageal disease with second-generation capsule endoscopy: initial evaluation of the PillCam ESO 2. Endoscopy. 2008 Apr;40(4):275-9. doi: 10.1055/s-2007-995645. PMID 18389444
- See also: Feasibility and Safety of magnetically controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3655386/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients over the age of 18 years old who required an EGD evaluation as part of a standard evaluation of relevant symptoms were approached regarding their willingness to have an MCCE examination. Patients needed to have one of several standard indicators for EGD, and none of the exclusion criteria. Additionally, patients planning on receiving a magnetic resonance imaging exam in the following 30 days were excluded. The study period lasted between February 10, 2021 and June 10, 2022.
Pre-assignment Details: There weren't any significant events following participant enrollment, but prior to assignment of participants to an arm or group.
Groups:
- MCCE(Magnetically Controlled Capsule Endoscopy) & EGD: In this prospective, single-arm, single-center, comparative study, adult patients aged ≥18 years who were referred for an EGD as part of a standard evaluation for symptoms were approached for participation in the study. Participants received MCCE before the EGD. MCCE videos were reviewed by 2 independent physicians and compared with subsequent EGD. Patients were followed for 30 days for safety outcomes and satisfaction.
Period: Overall Study
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Started | 43
Completed | 40
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 18 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 18
  Race: White | 14
  Race: Asian | 1
  Race: Other Race | 7
Region of Enrollment [Number; unit: participants]
  United States | 40
Medical History [Number; unit: participants]
  Diabetes mellitus | 2
  Kidney failure or on dialysis | 1
  Previous smoker/active smoker | 1
  Ulcer, gastritis, or acid reflux | 3
  Hemorrhoids | 1
  Other | 17
  None | 15
Medications [Number; unit: participants]
  Proton pump inhibitors | 15
  Nonsteroidal anti-inflammatory drugs | 7
Reasons for EGD Referral [Number; unit: participants] — Participants could have been referred for more than one reason
  participants
    Low blood (unexplained anemia) | 5
    Upper abdominal or chest pain | 15
    Indigestion (dyspepsia) | 3
    GERD | 9
    Suspected ulcer | 2
    Melena | 2
    Other | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Visualization of All Major Anatomic Regions in the Stomach With MCCE Based on 2 Reviewers
Description: Show that MCCE can identify anatomic regions of stomach consistent with established quality metrics for traditional endoscopy (>90% photo-documentation of pre-established anatomic regions). Each of the 40 MCCE results were reviewed by at least 2 physician reviewers for their ability to document the lower esophagus, Gastroesophageal junction/Z-line, and 6 gastric landmarks the cardia, fundus, body, angularis, antrum, and pylorus.
Time Frame: 90min
Measure: Number; unit: participants
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Number analyzed (Participants) | 40
participants
  Physician Reviewer 1 : No. of cases Cardia was visualized | 37
  Physician Reviewer 1 : No. of cases Fundus was visualized | 39
  Physician Reviewer 1 : No. of cases Body was visualized | 39
  Physician Reviewer 1 : No. of cases Angularis was visualized | 36
  Physician Reviewer 1 : No. of cases Antrum was visualized | 38
  Physician Reviewer 1 : No. of cases Pylorus was visualized | 39
  Physician Reviewer 1 : No. of cases Lower esophagus was visualized | 39
  Physician Reviewer 1 : No. of cases gastroesophageal junction/Z-line was visualized | 31
  Physician Reviewer 2 : No. of cases Cardia was visualized | 39
  Physician Reviewer 2 : No. of cases Fundus was visualized | 36
  Physician Reviewer 2 : No. of cases Body was visualized | 39
  Physician Reviewer 2 : No. of cases Angularis was visualized | 39
  Physician Reviewer 2 : No. of cases Antrum was visualized | 39
  Physician Reviewer 2 : No. of cases Pylorus was visualized | 39
  Physician Reviewer 2 : No. of cases Lower esophagus was visualized | 39
  Physician Reviewer 2 : No. of cases gastroesophageal junction/Z-line was visualized | 34

2. Primary Outcome: Comparison to EGD in Identifying Lesions.
Description: The goal of this assessment was to show that MCC is non-inferior to EGD in detecting both anatomic regions and gastric mucosal lesions
Time Frame: 5 Days
Measure: Count of Participants; unit: Participants
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Number analyzed (Participants) | 40
Participants
  no high-risk lesions were missed with MCCE | 35
  patients did not receive a follow-up EGD | 5

3. Secondary Outcome: Patient Preference Compared to EGD
Description: Measure patient preference for EGD vs MCC with a questionnaire. This will be used to document patient satisfaction from the ingestion of capsule to the 30 day follow-up period.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Number analyzed (Participants) | 40
Participants
  Patients preferred MCCE | 31
  Patients preferred EGD | 3
  Patients had no preference | 5
  Patients did not answer the question | 1

4. Secondary Outcome: Safety of MCC Compared to EGD. Documentation of Any Adverse Event Patient Encounters up to the 30 Day Follow-up.
Description: Measure the adverse events after MCC. This will be assessed using a questionnaire which will document any adverse event patient encounters up to the 30 day follow-up.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
Number analyzed (Participants) | 40
Participants
  No adverse outcome reported | 39
  Adverse outcome reported | 0
  Did not respond | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the day of study enrollment until the 30 day follow up call.
Description: Definition does not differ from clinicaltrials.gov
Arm/Group | MCCE(Magnetically Controlled Capsule Endoscopy) & EGD
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Limitation of the study included its small sample size and low number of pathologic lesions. In addition, although the GI endoscopist was blinded to the findings of the MCCE, the second physician interpreting the MCCE (physician reviewer 2) was not blinded to the interpretation of the initial MCCE operator (physician reviewer 1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04724291/Prot_000.pdf
  • Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT04724291/ICF_001.pdf